CLINICAL TRIAL: NCT04251065
Title: A Phase II, Open Label, Multicenter Trial of Daratumumab in Combination With Gemcitabine, Dexamethasone and Cisplatin (D-GDP) in Patients With Relapsed/Refractory CD38 Positive Peripheral T-cell Lymphoma Not Otherwise Specified (PTCL-NOS), Angioimmunoblastic T-cell Lymphoma (AITL) and Other Nodal Lymphomas of TFH Cell Origin
Brief Title: Daratumumab Plus Gemcitabine, Dexamethasone, Cisplatin in pt R/R CD38+ PTCL-NOS, AITL and TFH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrolment was prematurely terminated after the planned monitoring of the first 5 patients because of an unacceptable level of relevant toxicities, according to statistical stopping rules and the DSMB recommendation.
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_Dara-GDP
Record Dates: First submitted 2020-01-10; First posted 2020-01-31 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2022-11

CONDITIONS: Refractory T-Cell Lymphoma; Relapsed T-Cell Lymphoma
Keywords: CD38 positive; R/R peripheral T-cell lymphoma (PTCL-NOS); R/R angioimmunoblastic T-cell lymphoma (AITL); R/R nodal lymphomas of T follicular helper (TFH) cells; Daratumumab; Gemcitabine; Dexamethasone; Cisplatin
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single arm, single-stage phase II trial in patients with refractory/relapsed CD38 positive PTCL-NOS, AITL and TFH with centrally assessed CD38 expression ≥ 5%.
  It is expected for the current trial that D-GDP will improve the CR rate to 40% with an absolute improvement of 20%, while the toxicity rate is maintained at 30%.
  Sample size: A'Hern's Single-Stage Phase II design will be used. The sample size was calculated according to the primary efficacy endpoint. Based on literature, the null hypothesis that the true proportion of CR after four courses of D-GDP is 0.20 will be tested against an alternative CR proportion of 0.40 with an absolute improvement of 0.20, considered clinically promising with the experimental treatment. Assuming a type I error rate of 5% and a power of 80% when the CR proportion is 40% overall 35 patients will be accrued. The null hypothesis will be rejected if 12 or more CR out of 35 patients are observed after four courses of D-GDP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab-GDP (Experimental): This is an open-label, multicenter, single arm, single-stage phase II trial. After the patient signs the written informed consent the patient will enter the screening phase planning baseline assessments and a concomitant upfront confirmation of diagnosis of PTCL-NOS, AITL or nodal lymphoma of TFH cell origin and a central evaluation of immunohistochemical positivity of CD38 on bioptic material used to perform local diagnosis of relapsed disease, or that used for the more recent biopsy in the case of refractory patients. A core needle biopsy is considered sufficient for review and CD38 evaluation. Evaluation at central laboratory can be performed in bone marrow sections in those patients with only bone marrow lymphoma infiltration.
  Only patients with confirmed eligible diagnosis and a percentage of CD38 positive tumor cells ≥ 5% will be considered eligible for study treatment.
  The treatment consists of an induction phase and a maintenance phase.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab in combination with Gemcitabine, Dexamethasone and Cisplatin (D-GDP).
  Induction phase:
  4-6 courses (according to response after cycle 4 and to patient compliance) of D-GDP every 21 days pursuant to the following schedule: Daratumumab cycle 1: 8 mg/kg i.v. on day 2 and on day 9; cycle 2-6: 16 mg/kg i.v. on day 2 and day 9) Gemcitabine 1000 mg/sm i.v. day 1 and day 8 (gemcitabine on day 8 to be skipped in case of grade 3-4 toxicity) Cisplatin 75 mg/sm i.v. day 1 Dexamethasone 40 mg i.v. or po days 1-2-3-4-9 G-CSF from day 3 to 6, and from day 10 to 13 (to be prolonged if necessary)
  Maintenance:
  starting 28 days after the beginning of cycle 4 or 6 (or, in case of toxicity grade > 1, after toxicity is resolved) and up to 24 cycles from start of D-GDP according to the following schedule: Daratumumab 16 mg/kg single administration every 28 days.
  Other Names: Darzalex

SUMMARY:
FIL_Dara-GDP is a phase II, open label, multicenter clinical trial. The sponsor of this clinical trial is Fondazione Italiana Linfomi (FIL). The primary objective is to evaluate the efficacy of 4 courses of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) in terms of complete response in patients with peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL) and other nodal lymphomas of T follicular helper cells (TFH cells) origin refractory/relapsed after at least one and no more than two previous lines of therapy.

DETAILED DESCRIPTION:
This is an open-label, multicenter, single arm, single-stage phase II trial. After the patient signs the written informed consent the patient will enter the screening phase planning baseline assessments and a concomitant upfront confirmation of diagnosis of Peripheral T-Cell Lymphoma Not Otherwise Specified (PTCL-NOS), Angioimmunoblastic T-cell lymphoma (AITL) or Nodal Lymphoma of T Follicular Helper cells (TFH cells) origin and a central evaluation of immunohistochemical positivity of CD38 (cluster of differentiation 38) on bioptic material used to perform local diagnosis of relapsed disease, or that used for the more recent biopsy in the case of refractory patients. A core needle biopsy is considered sufficient for review and CD38 evaluation. Evaluation at central laboratory can be performed in bone marrow sections in those patients with only bone marrow lymphoma infiltration.

Only patients with confirmed eligible diagnosis and a percentage of CD38 positive tumor cells ≥ 5% will be considered eligible for study treatment.

The treatment consists of an induction phase and a maintenance phase.

Induction phase:

4-6 courses (according to response after cycle 4 and to patient compliance) of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) every 21 days pursuant to the following schedule:

* Daratumumab cycle 1: 8 mg/kg i.v. on day 2 and on day 9; cycle 2-6: 16 mg/kg i.v. on day 2 and day 9)
* Gemcitabine 1000 mg/sm i.v. day 1 and day 8 (gemcitabine on day 8 to be skipped in case of grade 3-4 toxicity)
* Cisplatin 75 mg/sm i.v. day 1
* Dexamethasone 40 mg i.v. or po days 1-2-3-4-9
* Granulocyte-colony stimulating factor (G-CSF) from day 3 to 6, and from day 10 to 13 (to be prolonged if necessary) After 4 courses of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone), patients in Complete Remission/Partial Remission (CR/PR) and eligible for allogeneic stem cell transplantation (allo-SCT) will be addressed to allo-SCT consolidation.

Otherwise, patients in Complete Remission (CR) will enter the maintenance phase at this point of the study.

Patients in Partial Remission (PR) (not eligible for allogeneic stem cell transplantation) or in Stable Disease (SD) after D-GDP x 4 cycles can receive 2 additional courses of D-GDP before maintenance or can move directly to maintenance, according to center choice (based on patient condition, performance status and quality of response).

Patients who respond (Complete Remission/Partial Remission) after 6 courses of induction phase (end of induction, EOI) and eligible to allogeneic stem cell transplantation (allo-SCT) will be addressed to allo-SCT consolidation.

Patients who respond to the induction phase (Complete Remission/Partial Remission) and are not eligible for allogeneic stem cell transplantation (allo-SCT) and patients in stable disease (SD) at the End Of Induction (EOI), will move to the maintenance phase.

Patients in Progressive disease (PD) at any time will discontinue treatment, as well as patients experiencing at any time unacceptable toxicity.

Maintenance phase:

starting 28 days after the beginning of cycle 4 or 6 (or, in case of toxicity grade > 1, after toxicity is resolved) and up to 24 cycles from start of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) according to the following schedule:

• Daratumumab 16 mg/kg single administration every 28 days

Treatment with D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) or daratumumab single agent will be discontinued before completion of 24 cycles in case of:

* decision of the investigator to consolidate D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) response with allogeneic stem cell transplant
* disease progression
* unacceptable toxicity
* withdrawal of consent
* investigator determines that further therapy is not in the patient's best interest (e.g., due to non-compliance, toxicity, etc.) Adverse events ("Common Terminology Criteria for Adverse Events", CTCAE v. 5.0) will be monitored from the first study-related procedure, throughout treatment, maintenance and for 30 days after the end of treatment with the study drug.

Safety monitoring and stopping rules:

In order to monitor the safety and the activity of the treatment in small cohorts of patients, the Bayesian approach of Thall et al. (1995), as extended by Thall and Sung (1998) will be used.

Monitoring of relevant toxicity after 4 cycles of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) will be done to ensure that it is not higher than an acceptable toxicity of 30% (as defined in the safety endpoints) and the monitoring of activity after 4 cycles of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) will be done to ensure that Complete Remission (CR) proportion is not lower than 40%.

The prior probability of toxicity and activity are modeled by beta distributions [Beta (0.6,1.4) and Beta (0.8,1.2), respectively].

The enrolment will be stopped if the posterior probability of the treatment being more toxic or less active than expected is greater than 95%.

The primary efficacy analysis will be performed after enrolment of 35 patients. The primary efficacy analysis will consist of an estimate of Complete Remission Rate (CRR) on the efficacy population after 4 cycles of D-GDP (Daratumumab in combination with Gemcitabine, Cisplatin, Dexamethasone) therapy, with 90% confidence intervals (according to 1-sided alpha error of 0.05). To conclude that the new treatment is promising, the minimum number of patients with a Complete Remission (CR) is 12/35.

The time-to-event functions (Overall Survival (OS) and Progression Free Survival (PFS)) will be estimated by the Kaplan-Meier product-limit method.

Subgroup analyses on primary efficacy parameter (Complete Remission Rate (CRR)) will be performed to assess the role of daratumumab maintenance and to explore potential prognostic role of CD38 expression. A logistic regression model will be used and the effect (Complete Remission Rate (CRR)) and its 95% Interval of Confidence (CI) will be presented.

For safety analysis, both at patient level and at therapy cycle level, summaries of incidence rates (frequencies and percentages) and intensity of individual adverse events by CTCAE (Common Terminology Criteria for Adverse Events (CTCAE)) v. 5.0 will be reported.

The results of this study will support the rationale of a phase III randomized trial if both efficacy and safety endpoints will be considered promising.

ELIGIBILITY:
Inclusion Criteria:

• Histologically documented diagnosis of CD38 (cluster of differentiation 38) positive PTCL-NOS, AITL and other nodal lymphomas of TFH cell origin as defined in the 2017 edition of the World Health Organization (WHO) classification. Patients with only bone marrow involvement are eligible.

Note: Only patients with a centrally assessed percentage of CD38 positive tumor cells ≥ 5% in the relapse biopsy, or in the more recent biopsy in the case of refractory patients, will be considered eligible for protocol study treatment.

* Age 18-70 years
* Relapsed or refractory to one previous lines of treatment (autologous transplantation as a consolidation to the first line of therapy should not be considered a second line)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) < 2
* At least one site of measurable nodal disease at baseline ≥ 2.0 cm in the longest transverse diameter as determined by CT scan (MRI is allowed only if CT scan cannot be performed). Note: Patients with only bone marrow involvement are eligible
* Adequate hematological counts defined as follows:

  * Absolute Neutrophil count (ANC) > 1.0 x 109/L unless due to bone marrow involvement by lymphoma
  * Platelet count > 100.000/mm3 unless due to bone marrow involvement by lymphoma
* Adequate renal function defined as follows:

  - Creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)
* Adequate hepatic function per local laboratory reference range as follows:

  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN)
  * Bilirubin ≤1.5 x upper limit of normal (ULN)(unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Subject understands and voluntarily signs an informed consent form approved by an Independent Ethics Committee (IEC), prior to the initiation of any screening or study-specific procedures
* Subject must be able to adhere to the study visit schedule and other protocol requirements
* Life expectancy ≥ 3 months
* Women must be:

  * postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months)
  * surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
  * completely abstinent (periodic abstinence from intercourse is not permitted) or if sexually active, be practicing two highly effective methods of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double barrier method (e.g.: condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization) as local regulations permit, before entry, and must agree to continue to use the same method of contraception throughout the study. They must also be prepared to continue birth control measures for at least 3 months after terminating treatment.
  * Women of childbearing potential must have a negative pregnancy test at screening
* Men must agree to use an acceptable method of contraception (for themselves or female partners as listed above) for the duration of the study. Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Male even if surgically sterilized (i.e., status post vasectomy) must agree to 1 of the following:

  * practice effective barrier contraception during the entire study treatment period and through 3 months after the last dose of study drug, or
  * agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner] and withdrawal are not acceptable methods of contraception)

Exclusion Criteria:

* Histological diagnosis different from CD38 positive PTCL-NOS, AITL, and other nodal lymphomas of TFH cell origin
* More than two lines of previous treatment (autologous stem cell transplant performed as part of consolidation to a previous line of therapy should not be considered as a line of therapy)
* Previous treatment with Gemcitabine or Platinum based regimens; patients who received a single course of Platinum based course (i.e. DHAP) are not excluded
* Prior therapy with monoclonal antibody anti CD38 (against cluster of differentiation 38)
* Concomitant experimental therapy
* Relapse after allo SCT
* Central nervous system (CNS) involvement with lymphoma
* Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, investigational therapy, including targeted small molecule agents within 14 days prior to the first dose of study drug
* Chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring treatment
* Subject is:

  * Known to be seropositive for human immunodeficiency virus (HIV)
  * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-hepatitis B core antigen (HBc)] ± antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
  * Known to be seropositive for hepatitis C (except in the setting of a Sustained Virologic Response(SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Cardiovascular disease (NYHA class ≥2)
* Creatinine Clearance < 40 mL/min (Cockcroft-Gault formula)
* Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent
* Any history of other active malignancies within 3 years prior to study entry, with the exception of adequately treated in situ carcinoma of the cervix uterine, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically resected with curative intent.
* Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
* Evidence of any other clinically significant uncontrolled condition(s)
* If female, the patient is pregnant or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Principal Investigator — S.C. Ematologia, Trieste - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia
Locations (7):
- Italy (7):
  - IRCCS Istituto Tumori Giovanni Paolo II - U.O.C Ematologia, Bari
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Ematologia, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - Trieste - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study stopped after the enrollment of 8 patients over the planned 35.
Groups:
- One Arm: Daratumumab in combination with Gemcitabine, Dexamethasone and Cisplatin (D-GDP) in patients with relapsed/refractory CD38 positive peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL) and other nodal lymphomas of TFH cell origin.
Period: Overall Study
Arm/Group | One Arm
Started | 8
Completed | 2
Not Completed | 6
Not completed — Death | 2
Not completed — Lack of Efficacy | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | One Arm
Number analyzed (Participants) | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [62.0 to 72.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Disease status at study entry [Count of Participants; unit: Participants]
  Relapse | 5
  Refractory | 3
Systemic B symptoms [Count of Participants; unit: Participants] — Symptoms B: absence of systemic symptoms; systemic symptoms defined as Night sweating, fever or Weight loss.
  Participants
    Absent | 4
    Present | 4
Ann Arbor Stage [Count of Participants; unit: Participants] — Staging for lymphomas disease, ranging from I (disease located in single region) to IV (diffuse or disseminated involvement of one or more extralymphatic organs)
  Participants
    III | 1
    IV | 7
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance status: scale ranging from 0 (person fully active) to 5 (death)
  Participants
    0 | 4
    1 | 4
Bone marrow involvement [Count of Participants; unit: Participants]
  Negative | 4
  Positive | 4
Number extra-nodal sites [Count of Participants; unit: Participants] — Extranodal localization by CT scan or combined PET-CT (Magnetic Resonance Imaging if CT cannot be done).
  Participants
    1 | 2
    2 | 2
    3 | 2
    4 | 1
    5 | 1
Type of the 1st Line Treatment [Count of Participants; unit: Participants] — CHOEP: cyclophosphamide doxorubicin vincristine Etoposide Prednisone DHAP: rituximab dexamethasone cytarabine cisplatin ASCT: autologous stem cell transplant ARA-C: cytarabine CHOP: cyclophosphamide doxorubicine vincristine prednisone COEP: cyclophosphamide etoposide vincristine prednisone HSCT: haematopoietic stem cell transplantation
  Participants
    6 cy CHOEP + 1 cy DHAP + ASCT | 1
    6 cy CHOP+DHAP+ASCT | 2
    CHOEP | 1
    6cy CHOEP + ARA-C + ABMT | 1
    CHOP | 1
    COEP | 1
    CHOEP +HSCT | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR)
Description: The Complete Response Rate is defined as the percentage of patient in Complete Remission (according to Lugano classification response Criteria). It will be assessed after the first 4 cycles of D-GDP chemotherapy. In case of early discontinuation, efficacy will be assessed at the End Of Treatment (EOT) visit. Patients without response assessment (due to whatever reason) will be considered as non-responders. CR: complete radiological response, no extralymphatic sites, no new lesions, organ enlargement regress to normal and normal morphology of bone marrow; PR: >=50% decrease of sum of the product of perpendicular diameter of up to 6 dominant, measurable nodes and and extranodal sites.
Time Frame: the endpoint will be assessed from the start date of therapy to the end of the first four cycles of therapy (cycles of 21 days).
Measure: Count of Participants; unit: Participants
Arm/Group | One Arm
Number analyzed (Participants) | 8
Participants
  CRR | 0
  Less than CRR | 8

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate is defined as the percentage of patients in complete remission or in partial remission (according to the Lugano 2014 criteria) after the first 4 cycles of therapy (cycles of 21 days). Patients without response assessment (due to whatever reason) will be considered as non-responders. CR: complete radiological response, no extralymphatic sites, no new lesions, organ enlargement regress to normal and normal morphology of bone marrow; PR: >=50% decrease of sum of the product of perpendicular diameter of up to 6 dominant, measurable nodes and and extranodal sites.
Time Frame: the endpoint will be assessed from the start date of therapy to the end of the first four cycles of therapy (cycles of 21 days) and at each restaging
Measure: Count of Participants; unit: Participants
Arm/Group | One Arm
Number analyzed (Participants) | 8
Participants
  ORR | 1
  Less than ORR | 7

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival, the percentage of patients alive, is defined from the start date of therapy to the date of death from any cause. Patients alive and those who are lost to follow-up at the time of the final analysis will be censored at the date of the last contact.
Time Frame: The end point will be assessed from the start date of therapy up to 3 months.
Measure: Number (95% Confidence Interval); unit: Percent probability at 3 months
Arm/Group | One Arm
Number analyzed (Participants) | 8
Percent probability at 3 months | 62.5 [22.9 to 86.1]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: The length of time during and after the treatment that patients live with the disease, but it does not get worse. Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.
  Responding patients, according to the Lugano classification response Criteria, and patients who are lost to follow-up will be censored at their last assessment date.
Time Frame: The endpoint will be assessed from the start date of therapy up to 3 months.
Measure: Number (95% Confidence Interval); unit: Percent probability at 3 months
Arm/Group | One Arm
Number analyzed (Participants) | 8
Percent probability at 3 months | 50.0 [15.2 to 77.5]

5. Secondary Outcome: Toxicity - Frequency of Relevant Toxicities
Description: Frequency of relevant toxicities. Toxicities will be classified according to Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. This endpoint will be evaluated from the start date of therapy and at any time during therapy and follow-up.
Time Frame: the endpoint was assessed after 26 months from the date of starting therapy in place of the planned 42 months, due the early interruption of the study
Population: Monitoring planned after the first 5 patients treated.
Measure: Count of Participants; unit: Participants
Arm/Group | One Arm
Number analyzed (Participants) | 5
Participants
  Septic shock multi-organ failure | 1
  Acute myocardial infraction | 1
  Thrombocytopenia | 2
  No relevant event | 1

6. Other Pre Specified Outcome: Role of Daratumumab Maintenance
Description: Comparison between the Complete Remission Rate (CRR), percentage of patient in complete remission, before and after maintenance therapy
Time Frame: The endpoint will be assessed at each restaging through study completion, up to 26 months.
Population: Due the early interruption of the trial, this end point was not evaluated.
Arm/Group | One Arm
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Role of Daratumumab Maintenance CR vs PR
Description: The evaluation of the rate of conversion in Complete Remission with daratumumab maintenance therapy for patients in Partial Remission after the induction.
  With this endpoint it will be measured the number of responses that will be converted from Partial Remission (PR) to Complete Remission (CR) in those patients that after induction therapy continued the treatment with the maintenance therapy.
Time Frame: The endpoint will be assessed at each restaging through study completion, up to 26 months.
Population: Due the early interruption of the trial, this end point was not evaluated. So, data were not collected.
Arm/Group | One Arm
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Percentage of CD38 Expression in Correlation With the Response to the Treatment
Description: This endpoint will evaluate the correlation between intensity of CD38 expression (percentage of expression) and response to the treatment. The extent of CD38 expression evaluated by the central designed laboratory of FIL (Fondazione Italiana Linfomi) will be performed on fresh sections cut from the paraffin block (or on unstained sections), and the percentage of positive tumor cells will be scored according to Bossard C. et al as follows: 4: >75%; 3: 50-75%; 2: 25-49%; 1: 5-24%; 0: <5%. The percentage of CD38 expression will be correlated with response measured according to the Lugano 2014 criteria
Time Frame: The endpoint will be assessed from the start date of therapy to the end of the first four cycle of therapy (cycles of 21 days) and at each restaging through study completion, up to 26 months.
Population: No data displayed because Outcome Measure has zero total participants analyzed. So, data were not collected.
Arm/Group | One Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The endpoint was assessed after 26 months from the date of starting therapy in place of the planned 42 months, due the early interruption of the study
Description: CTCAE
Arm/Group | One Arm
All-Cause Mortality (participants affected / at risk) | 8/8
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Arm (N=8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
septic shock multiorgan failure (Infections and infestations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1)
Thenth rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
EBV infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Arm (N=8)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
General disorder (General disorders) | 4 (4)
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (1)
Immuno system (Immune system disorders) | 1 (1)
Infections (Infections and infestations) | 4 (4)
Investigations (Investigations) | 1 (1)
Metabolism (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal and urinary (Renal and urinary disorders) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Other (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Due early termination, only 8 patients were enrolled in the study. The study highlight a high level of toxicity of the experimental treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT04251065/Prot_SAP_000.pdf